CLINICAL TRIAL: NCT06430138
Title: Bioavailability and Bioactivity of Orange Polyphenols on Gut Health
Brief Title: Bioavailability and Bioactivity of Orange Polyphenols
Acronym: ORANGUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Andalusian Institute of Agricultural and Fisheries Research and Training (IFAPA) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: REC/24/0002
Record Dates: First submitted 2024-04-23; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-04

CONDITIONS: Healthy Nutrition
Keywords: Orange,; polyphenols; ileostomy

STUDY DESIGN:
Intervention Model Description: Acute intervention in populations with and without colon
Who Masked: Participant
Masking Description: Single Blind(with masked participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy participants (Experimental): Participant will be given Orange Juice 300ml to drink
  Interventions: Dietary Supplement: 300ml Orange Juice
- Ileostomy participants (Active Comparator): Participant will be given orange Juice 300ml to drink
  Interventions: Dietary Supplement: 300ml Orange Juice

INTERVENTIONS:
Dietary Supplement: 300ml Orange Juice — Acute intervention in populations with and without colon

SUMMARY:
This study will provide a greater insight into the relationship between orange consumption and health (particularly gut health) and could be used to help with the development of novel food products. Oranges are a rich source of (poly)phenols, and although the advantages of a (poly)phenol-rich diet are well-established, the bioavailability and bioactivity of orange (poly)phenols in the context of human digestion are poorly understood. This study will address this gap in research.

DETAILED DESCRIPTION:
This study will provide a greater insight into the relationship between orange consumption and health (particularly gut health) and could be used to help with the development of novel food products. Oranges are a rich source of (poly)phenols, and although the advantages of a (poly)phenol-rich diet are well-established, the bioavailability and bioactivity of orange (poly)phenols in the context of human digestion are poorly understood.

Until recently, analysis of biofluids with HPLC-MS revealed relatively simple phenolic profiles. However, with current high resolution (HR)-MS instrumentation detection limits and selectivity have improved greatly and HPLC-HR-MS methodology is now the analytical method of choice. Consequently, the number of phenolics that can be monitored has increased markedly in recent years. A previous study, using validated methodology, identified 65 phenolic compounds in urine collected after ingestion of orange juice.

In the proposed project it is planned to use such analytical methodology for targeted and untargeted metabolomics of flavanone metabolites and colonic catabolites in biofluids collected after consumption of orange juice by ileostomists and subjects with a functioning colon. Metabolomics refers to the measurement of metabolites present within a cell, tissue, or organism resulting from physiological stimulus - in the context of the current study, the stimulus is orange juice consumption. Untargeted metabolomics involves a comprehensive analysis of all measurable substances in a sample of unknown metabolites, and targeted metabolomics denotes the quantification of defined group(s) of metabolites. The particular value of including ileostomists in the study is that analysis of their ileal fluid and urine will provide valuable information on compounds derived from the ingested OJ flavanones, prior to digestion and absorption by the large intestine.

Acute bioavailability feeding study in two groups; ileostomists and healthy adults. The study will take place in the Human Intervention Studies Unit (HISU), at Ulster University, Coleraine Campus. Prior to attending the HISU, participants will be asked to follow a restriction diet for 72 hours before the study and the 24 hours of the study day, which will involve the intake of food containing low levels of (poly)phenols. The participants will be provided with a restriction (low (poly)phenol) meal, which they will consume the evening before the study (at approximately 6 - 7.00pm) and fast until attending the HISU the following morning. This means no food will be taken overnight and no breakfast taken prior to attending the HISU.

Low (poly)phenol foods will be provided to participants on the day of the study, and they will be asked to continue this restriction diet until all samples have been collected. Healthy participants and Ileostomists (N=20) will provide 10 blood samples and 3 urine samples over the study period.

Blood samples:

Upon arrival at the HISU, a qualified phlebotomist will fit a cannula, and collect a blood sample (0hr) (~8ml). The participant will then be given the intervention; 300 ml of orange juice. A further 8 blood samples will be collected at 1hr intervals (1hr, 2hr, 3hr, 4hr, 5hr, 6hr, 7hr, 8hr). After the 8hr blood draw the cannula will be removed by the phlebotomist and the participant will be free to go home. They will return to the HISU the following morning to provide a final blood sample (24hr). Ten blood samples will be collected in total.

Urine samples:

Participants will start a 24-hour urine collection the day before the study day. They will be provided with a 2L urine container in advance of commencing the urine collection; participants will use this to deposit urine samples over the 24-hr period. Upon arrival at the HISU on the morning of the study, participants will return the urine container holding the -24 to 0 hr urine sample. Participants will complete two additional urine collections (0-8hr and 8-24hr samples), a fresh urine container will be provided at each time point. The 8-24hr sample will be returned by the participant when they return to the HISU to provide the 24hr blood sample.

Ileostomist participants (n=10) will also provide three ileal samples over the study period.

Ileal samples:

Participants will be asked to refrain from emptying their stoma bag upon waking on the morning of the study. Upon arrival at the HISU, an ileal sample will be collected; the overnight stoma bag will be removed and replaced with a new stoma bag by the participant. Two additional ileal samples will be collected at 0-8 hr and 8-24 hrs, the stoma bag will be removed and replaced with a new stoma bag by the participant at each sampling point. The 8-24hr sample will be returned by the participant when they return to the HISU to provide the 24hr blood sample. Multiple stoma bags may be used by the participant as required.

Height and weight measurements will also be taken for all participants (N=20), during their visit to the HISU.

ELIGIBILITY:
Inclusion Criteria: (ileostomates)

* Adult with an ileostomy, ≥1.5-years post-operative
* Aged 18-75 years at recruitment
* Not pregnant / lactating
* No learning or other disabilities
* Not currently taking antibiotics
* Not currently taking plant-based dietary supplements
* Not currently taking any prescribed medications that would prevent overnight fasting

Inclusion Criteria Healthy adults; no pre-existing chronic disease (GI related)

* Aged 18-75 years at recruitment
* Not pregnant / lactating
* No learning or other disabilities
* Not currently taking antibiotics
* Not currently taking plant-based dietary supplements
* Not currently taking any prescribed medications that would prevent overnight fasting

Exclusion criteria (Ileostomates):

* Adults <18 or >75 years at recruitment
* Ileostomy, <1.5 years post-operative
* Pregnant/lactating females
* Adults with learning or other disabilities
* Citrus fruit (orange) allergy or sensitivity
* Currently taking antibiotics
* Currently taking plant-based dietary supplements
* Currently taking any prescribed medications that would prevent overnight fasting

Exclusion criteria (Healthy adults):

* Adults <18 or >70 years at recruitment
* Pregnant/lactating females
* Adults with learning or other disabilities
* Citrus fruit (orange) allergy or sensitivity
* Currently taking antibiotics
* Currently taking plant-based dietary supplements
* Currently taking any prescribed medications that would prevent overnight fasting

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-09-13 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Quantification of circulating (blood) (poly)phenols and microbially derived metabolites in participants with colon compared to without colon (ileostomates). | Change over 24 hours compared
  Quantification of polyphenols via LC-MS/MS
Quantification of urinary (poly)phenols and microbially derived metabolites in participants with colon compared to without colon (ileostomates). | Change over 24 hours ]
  Quantification of polyphenols via LC-MS/MS

SECONDARY OUTCOMES:
ileal fluid polyphenolic metabolites. | Change over 24 hours
  Mass spectrometry analysis of In vitro gut model colonic fermentation of ileal fluid (µmol/L)
Ileal fluid microbial mediated metabolites | Change over 24 hours
  Mass spectrometry analysis of In vitro gut model colonic fermentation of ileal fluid (µmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Ulster University,Human Intervention Studies Unit,, Coleraine, Co. Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No